CLINICAL TRIAL: NCT00678652
Title: Ph 1 Dose-Escalation Study of Safety and Immunogenicity of 3 Injections, at 0, 6, 2 Wks, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine Adm Intramuscularly to Healthy Subjects at 10, 25, 50, 75 μg With Adjuvant
Brief Title: Phase 1 Safety and Immunogenicity of Meningococcal Vaccine
Acronym: HOPS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR 1395; HSRRB Log A-14553 (Other: IRB); MIDRP AM0035_07_WR (Other); S-15-08 (Other: Sponsor)
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Meningococcal Infection, Group B
Keywords: Meningococcal vaccine; Neisseria meningitidis
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine (Experimental): Three Injections, Given at 0, 6, and 12 Weeks, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine Administered Intramuscularly to Healthy Subjects at 10 μg with Adjuvant
  Interventions: Biological: 10 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine
- 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine (Experimental): Three Injections, Given at 0, 6, and 12 Weeks, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine Administered Intramuscularly to Healthy Subjects at 25 μg with Adjuvant
  Interventions: Biological: 25 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine
- 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine (Experimental): Three Injections, Given at 0, 6, and 12 Weeks, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine Administered Intramuscularly to Healthy Subjects at 50 μg with Adjuvant
  Interventions: Biological: 50 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine
- 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine (Experimental): Three Injections, Given at 0, 6, and 12 Weeks, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine Administered Intramuscularly to Healthy Subjects at 75 μg with Adjuvant
  Interventions: Biological: 75 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine

INTERVENTIONS:
Biological: 10 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine — 10 μg of Meningococcal 8570 HOPS-G NOMV Vaccine given at 0, 6, and 12 weeks, administered intramuscularly to healthy subjects for duration of study
  Arms: 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine
Biological: 25 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine — 25 μg of Meningococcal 8570 HOPS-G NOMV Vaccine given at 0, 6, and 12 weeks, administered intramuscularly to healthy subjects for duration of study
  Arms: 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine
Biological: 50 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine — 50 μg of Meningococcal 8570 HOPS-G NOMV Vaccine given at 0, 6, and 12 weeks, administered intramuscularly to healthy subjects for duration of study
  Arms: 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine
Biological: 75 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine — 75 μg of Meningococcal 8570 HOPS-G NOMV Vaccine given at 0, 6, and 12 weeks, administered intramuscularly to healthy subjects for duration of study
  Arms: 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine

SUMMARY:
The purpose of this study is to determine whether a vaccine based on outer membrane vesicles (NOMV) from genetically detoxified group B meningococcus is safe and effective for use as a vaccine. If so, the NOMV in this vaccine will be combined with NOMV from two other genetically modified strains as a potentially globally effective vaccine against group B meningococcus.

DETAILED DESCRIPTION:
This was a Phase 1, outpatient, open-label, dose-escalating study to evaluate the safety, tolerability, and immunogenicity of 4 doses of the Group B Meningococcal HOPS-G 8570 NOMV vaccine in healthy subjects. Subjects were screened by medical history; physical exam; complete blood count; serum chemistry profile; coagulation studies including prothrombin time (PT), partial thromboplastin time (PTT), and fibrinogen; human immunodeficiency virus (HIV) test, anti-hepatitis C virus (HCV) antibodies, and hepatitis B surface antigen (HBsAg) test results; nasopharyngeal swabs for carriage of meningococci; bactericidal antibody titer to meningococci; and urinalysis; and urine pregnancy test results for females. The first 36 subjects to meet all inclusion criteria and none of the exclusion criteria were assigned to 1 of 4 dosage groups of 9 subjects each. After screening, there was a 10 to 60 day lead-in time (depending on when screening occurred) prior to vaccination during which subjects could not take or receive any experimental products. Also prior to vaccination, adverse events were recorded to establish a baseline with which to compare adverse events occurring after vaccination. Subjects kept a diary for 7 days before the first dose and for 1 day before each of the second and third doses. Immediately before each vaccination, vital signs were checked, an abbreviated physical examination was performed, each subject's throat was swabbed to assess carriage of meningococcal bacteria, and blood was drawn for immunology and safety labs. Urine was collected for analysis and females took a urine pregnancy test. The pregnancy test results had to be negative in order for a subject to be vaccinated. The vaccine with adjuvant was given intramuscularly at 0, 6, and 12 weeks (Study Days 0, 42, and 84) in doses of 10 μg, 25 μg, 50 μg, or 75 μg based on protein concentration. Vaccinations were performed in a staggered fashion with safety monitoring between groups. The 10-μg dose group was divided into 2 subgroups. Subjects in the first subgroup were vaccinated 30 minutes apart to observe subjects for the occurrence of acute side effects, and subjects in the second subgroup were vaccinated 1 week after the first. The subjects in each group were monitored for AE for at least 2 weeks prior to vaccinating the next higher dosage group. Subjects were kept in the Clinical Trials Center for 30 minutes after each vaccination for observation, and they were asked to keep a diary of symptoms for 7 days after each vaccination. AEs and SAEs were recorded at all study visits, and each AE or SAE was assessed for severity and relationship to the vaccine by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (by physical examination and medical history) military or civilian males or females;
* Age 18-45 years;
* Able to give informed consent, understands risks and benefits of study, assents to use of blood samples for future research; understands and is willing to comply with all protocol procedures and time commitments;
* Females must have a negative urine pregnancy test on vaccination day before each dose AND agree to practice an effective birth control method as necessary, for 6 months after the first vaccination;
* Military service-members who wish to participate must obtain written permission from their immediate supervisor, department chief or equivalent, and company commander or equivalent.

Exclusion Criteria:

* Current or history of significant organ/system disease;
* History of allergy to any vaccine;
* History of allergy to aluminum hydroxide;
* Presence of significant unexplained laboratory abnormality that in the opinion of the PI may potentially confound the analysis of the study results;
* HIV seropositive or any other immunosuppressive state;
* Positive test for HBsAg or hepatitis C antibody;
* Evidence or admission of on-going drug or alcohol abuse/dependence;
* Intention to leave the area during the study such that the volunteer would miss 1 or more study days;
* Prior receipt of any group B meningococcal outer membrane protein (OMP) vaccine or a vaccine containing meningococcal OMP;
* Has received or plans to receive any live vaccine, Investigational New Drug (IND) products or significant immunosuppressive therapy* in the 28 days prior to, or any inactivated vaccine within 14 days before initial vaccination or throughout the study, or received parenteral immunoglobulin or blood products within 3 months of study initiation;

  * (Intra-articular, topical, or intranasal steroids, steroids applied to the eye, or ≤ 7 days of oral steroids are in general acceptable, depending on the formulation and condition for which they are prescribed. Inclusion of individuals receiving these medications will be made by the PI on a case by case basis)
* High levels of baseline bactericidal antibodies against the vaccine strain on screening (>1:16) and/or throat carriage of Neisseria meningitidis at time of screening;
* Positive urine pregnancy test prior to vaccination;
* Lactation from first dose through 3 months after last dose;
* Any condition in the opinion of the investigator that might interfere with the study vaccine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Keiser, M.D., Principal Investigator — WRAIR, Division of Bacterial and Rickettsial Diseases
Locations (1):
- Clinical Trials Center, WRAIR, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from CTC database if they have asked to be informed about upcoming studies. Posters//flyers, tv, internet, newspaper ads and word of mouth to recruit healthy subjects. Recruitment may include oral presentations and/or distribution of approved recruiting materials.
Groups:
- 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine: Three Injections, Given at 0, 6, and 12 Weeks, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine Administered Intramuscularly to Healthy Subjects at 10 μg with Adjuvant
  10 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine: 10 μg of vaccine given at 0, 6, and 12 weeks, administered intramuscularly to healthy subjects for duration of study
- 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine: Three Injections, Given at 0, 6, and 12 Weeks, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine Administered Intramuscularly to Healthy Subjects at 25 μg with Adjuvant
  25 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine: 25 μg of vaccine given at 0, 6, and 12 weeks, administered intramuscularly to healthy subjects for duration of study
- 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine: Three Injections, Given at 0, 6, and 12 Weeks, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine Administered Intramuscularly to Healthy Subjects at 50 μg with Adjuvant
  50 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine: 50 μg of vaccine given at 0, 6, and 12 weeks, administered intramuscularly to healthy subjects for duration of study
- 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine: Three Injections, Given at 0, 6, and 12 Weeks, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine Administered Intramuscularly to Healthy Subjects at 75 μg with Adjuvant
  75 μg Group B Meningococcal 8570 HOPS-G NOMV Vaccine: 75 μg of vaccine given at 0, 6, and 12 weeks, administered intramuscularly to healthy subjects for duration of study
Period: Overall Study
Arm/Group | 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine
Started | 9 | 9 | 9 | 9
Completed | 6 | 9 | 8 | 9
Not Completed | 3 | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Relocation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Customized [Count of Participants; unit: Participants] — 18 - 45 years old
  Participants
    18 - 45 | 9 | 9 | 9 | 9 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 4 | 14
  Male | 7 | 6 | 4 | 5 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 9 | 8 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 7 | 7 | 3 | 5 | 22
  White | 1 | 2 | 5 | 4 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Bactericidal Absolute Values After Group B Meningococcal 8570 HOPS-G NOMV Vaccine Injections
Description: Measure the bactericidal absolute values per dose group after vaccine injections, administered intramuscularly, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine at 10, 25, 50, or 75 μg with aluminum hydroxide adjuvant in healthy adult subjects.
Time Frame: 18 weeks. Days 0, 14, 56, 84, 98 and 126
Measure: Mean (Standard Deviation); unit: titers
Arm/Group | 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine
Number analyzed (Participants) | 7 | 9 | 9 | 9
titers
  Day 0 | 2.1 (1.5) | 3.0 (2.9) | 3.0 (2.3) | 2.4 (1.2)
  Day 14 | 7.0 (5.6) | 20.4 (21.1) | 12.4 (11.9) | 8.4 (9.2)
  Day 42 | 6.8 (5.8) | 13.1 (12.0) | 6.7 (5.6) | 5.3 (4.4)
  Day 56 | 5.0 (3.0) | 11.6 (9.6) | 8.9 (9.7) | 8.4 (9.2)
  Day 84 | 4.4 (2.7) | 10.9 (10.1) | 7.8 (5.5) | 6.9 (5.7)
  Day 98 | 8.0 (6.0) | 19.3 (12.9) | 11.6 (9.6) | 11.1 (9.1)
  Day 126 | 7.8 (6.8) | 10.2 (6.9) | 6.9 (4.7) | 6.0 (4.2)

2. Primary Outcome: Rate of Seroconversion After the 2nd Dose of 8570 L3-5,7-5 Vaccine
Description: Rate of seroconversion (fourfold increase from baseline in antibody titer of bactericidal antibodies) after the 2nd dose of vaccine
Time Frame: 42+7 days (visit 7)
Population: Seroconversion is defined as a 4-fold or greater increase from baseline in antibody titer of bactericidal antibodies after 2 doses (the first and second) of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine
Number analyzed (Participants) | 7 | 9 | 9 | 9
Participants
  Yes | 3 | 6 | 3 | 4
  No | 4 | 3 | 6 | 5

3. Primary Outcome: Rate of Seroconversion After the 3rd Dose of 8570 L3-5, 7-5 Vaccine
Description: Rate of seroconversion (fourfold increase from baseline in antibody titer of bactericidal antibodies) after the 3rd dose of vaccine
Time Frame: 84+7 days (visit 11)
Population: Seroconversion is defined as a 4-fold or greater increase from baseline in antibody titer of bactericidal antibodies after 3 doses of vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine
Number analyzed (Participants) | 7 | 9 | 9 | 9
Participants
  Yes | 5 | 8 | 5 | 6
  No | 2 | 1 | 4 | 3

4. Secondary Outcome: Total Antibody Response to the Parent Strain of Group B Meningococcus
Description: Assess and characterize bactericidal activity and total antibody response against the vaccine strain and other strains of Group B Meningococcus induced by 3 injections, administered intramuscularly, of Group B Meningococcal 8570 HOPS-G NOMV Vaccine at 10, 25, 50, or 75 μg with aluminum hydroxide adjuvant in healthy adult subjects.
Time Frame: 126 days
Measure: Median (Full Range); unit: ug/mL
Arm/Group | 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine
Number analyzed (Participants) | 9 | 9 | 9 | 9
ug/mL
  Antigen: GNA1870, Antibody Type: IgG - Day 0 | 3.4 [2.2 to 10.6] | 3.1 [0.9 to 7.2] | 2.7 [1.8 to 4.0] | 3.0 [0.8 to 4.0]
  Antigen: GNA1870, Antibody Type: IgG - Day 14 | 5.3 [1.8 to 13.3] | 3.3 [1.0 to 8.1] | 3.3 [2.1 to 10.2] | 3.9 [2.6 to 7.2]
  Antigen: GNA1870, Antibody Type: IgG - Day 56 | 4.2 [2.4 to 31.5] | 3.2 [2.6 to 8.4] | 3.4 [2.4 to 9.1] | 7.8 [3.0 to 12.2]
  Antigen: GNA1870, Antibody Type: IgG - Day 98 | 3.7 [2.5 to 29.2] | 3.9 [2.3 to 7.6] | 4.4 [2.8 to 11.1] | 11.6 [2.6 to 17.9]
  Antigen: L3, 7 LOS, Antibody Type: IgG - Day 0 | 0.4 [0.1 to 1.2] | 0.2 [0.1 to 0.3] | 0.3 [0.1 to 0.9] | 0.1 [0.1 to 0.5]
  Antigen: L3, 7 LOS, Antibody Type: IgG - Day 14 | 1.0 [0.1 to 2.3] | 0.3 [0.1 to 0.7] | 0.7 [0.2 to 1.8] | 0.7 [0.2 to 12.0]
  Antigen: L3, 7 LOS, Antibody Type: IgG - Day 56 | 0.7 [0.1 to 1.3] | 0.2 [0.1 to 0.4] | 0.6 [0.1 to 2.3] | 0.5 [0.2 to 3.7]
  Antigen: L3, 7 LOS, Antibody Type: IgG - Day 98 | 1.0 [0.2 to 2.3] | 0.3 [0.1 to 0.6] | 0.5 [0.1 to 2.6] | 1.1 [0.3 to 2.7]
  Antigen: L8-5 LOS, Antibody Type: IgG - Day 0 | 0.3 [0.1 to 0.8] | 0.1 [0.0 to 0.5] | 0.2 [0.1 to 2.7] | 0.1 [0.1 to 0.2]
  Antigen: L8-5 LOS, Antibody Type: IgG - Day 14 | 1.6 [0.3 to 10.8] | 0.6 [0.1 to 1.8] | 2.3 [0.4 to 3.8] | 1.9 [0.3 to 34.0]
  Antigen: L8-5 LOS, Antibody Type: IgG - Day 56 | 1.2 [0.4 to 2.9] | 0.5 [0.1 to 1.8] | 1.4 [0.3 to 3.7] | 1.3 [0.3 to 8.3]
  Antigen: L8-5 LOS, Antibody Type: IgG - Day 98 | 1.8 [0.7 to 5.7] | 0.7 [0.1 to 1.1] | 1.3 [0.2 to 3.1] | 2.5 [0.5 to 7.6]
  Antigen Type: OpeA, Antibody Type: IgG - Day 0 | 0.1 [0.0 to 0.3] | 0.1 [0.0 to 0.5] | 0.2 [0.0 to 1.1] | 0.1 [0.0 to 0.6]
  Antigen Type: OpeA, Antibody Type: IgG - Day 14 | 0.2 [0.1 to 0.5] | 0.1 [0.0 to 1.6] | 1.2 [0.1 to 7.4] | 0.2 [0.1 to 7.3]
  Antigen Type: OpeA, Antibody Type: IgG - Day 56 | 0.1 [0.1 to 0.4] | 0.2 [0.1 to 1.0] | 0.5 [0.1 to 3.6] | 0.2 [0.1 to 5.5]
  Antigen Type: OpeA, Antibody Type: IgG - Day 98 | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.8] | 0.5 [0.1 to 1.9] | 0.2 [0.1 to 1.6]
  Antigen: Vaccine NOMV, Antibody Type: IgG - Day 0 | 27.7 [4.7 to 58.3] | 13.2 [3.8 to 43.2] | 29.6 [11.5 to 52.7] | 13.8 [9.5 to 65.8]
  Antigen: Vaccine NOMV, Antibody Type: IgG - Day 14 | 50.8 [15.4 to 137.3] | 33.8 [8.9 to 160.8] | 74.3 [13.5 to 133.1] | 39.7 [17.2 to 189.6]
  Antigen: Vaccine NOMV, Antibody Type: IgG - Day 42 | 46.0 [16.3 to 91.8] | 23.4 [7.9 to 127.3] | 49.1 [19.1 to 84.6] | 24.2 [22.0 to 118.2]
  Antigen: Vaccine NOMV, Antibody Type: IgG - Day 56 | 62.7 [27.2 to 115.0] | 42.6 [10.9 to 129.4] | 44.4 [12.9 to 112.2] | 40.3 [22.1 to 205.7]
  Antigen: Vaccine NOMV, Antibody Type: IgG - Day 84 | 47.9 [20.7 to 102.1] | 29.4 [10.2 to 115.3] | 43.1 [12.6 to 114.1] | 33.4 [24.2 to 211.3]
  Antigen: Vaccine NOMV, Antibody Type: IgG - Day 98 | 51.3 [16.4 to 137.2] | 32.7 [11.8 to 119.8] | 45.3 [15.4 to 369.5] | 42.4 [27.8 to 208.6]
  Antigen: Vaccine NOMV, Antibody Type: IgG - Day126 | 50.7 [17.1 to 140.5] | 31.7 [14.1 to 129.3] | 45.6 [14.0 to 126.3] | 49.6 [21.7 to 164.0]
  Antigen: Vaccine NOMV, Antibody Type: IgM - Day 0 | 4.1 [2.4 to 10.7] | 7.8 [1.4 to 10.4] | 11.1 [2.7 to 14.1] | 3.8 [1.3 to 6.4]
  Antigen: Vaccine NOMV, Antibody Type: IgM - Day 14 | 6.3 [3.3 to 24.3] | 9.8 [2.1 to 41.9] | 14.2 [3.1 to 75.5] | 10.8 [2.6 to 40.2]
  Antigen: Vaccine NOMV, Antibody Type: IgM - Day 42 | 7.5 [2.8 to 14.0] | 9.9 [1.5 to 13.2] | 12.2 [3.1 to 14.2] | 7.4 [1.6 to 9.7]
  Antigen: Vaccine NOMV, Antibody Type: IgM - Day 56 | 10.4 [2.6 to 16.2] | 10.5 [1.8 to 12.8] | 11.7 [3.5 to 14.7] | 8.0 [1.9 to 11.7]
  Antigen: Vaccine NOMV, Antibody Type: IgM - Day 84 | 7.4 [3.0 to 10.8] | 8.6 [1.4 to 17.8] | 11.4 [3.2 to 15.7] | 7.1 [1.3 to 14.1]
  Antigen: Vaccine NOMV, Antibody Type: IgM - Day 98 | 9.8 [3.3 to 12.6] | 10.8 [1.7 to 14.7] | 10.7 [4.1 to 18.5] | 6.6 [2.8 to 14.1]
  Antigen: Vaccine NOMV, Antibody Type: IgM - Day126 | 8.2 [2.5 to 10.7] | 7.8 [1.6 to 14.3] | 10.5 [3.5 to 15.7] | 5.6 [2.0 to 11.3]

ADVERSE EVENTS:
Time Frame: 126 days +14
Arm/Group | 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine | 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 9/9 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine (N=9) | 25 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine (N=9) | 50 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine (N=9) | 75 μg of Group B Meningococcal 8570 HOPS-G NOMV Vaccine (N=9)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (5) | 3 (3) | 1 (1) | 2 (2)
Feeling Hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 8 (8) | 8 (8) | 8 (8) | 9 (9)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 5 (5) | 6 (6) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Asthenopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper Respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 5 (5) | 6 (6)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Excoriaton (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post concussoin syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Blood bicarbonate decreased (Investigations) | 4 (4) | 3 (3) | 8 (8) | 8 (8)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Blood fibrinogen decreased (Investigations) | 3 (3) | 5 (5) | 4 (4) | 1 (1)
Blood fibrinogen increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Blood glucose decreased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 5 (5)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blood pressure dastolic increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urine leukocyte esterase (Investigations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
White blood cell count increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraeshthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstrual discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis papillaris capillitii (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No